CLINICAL TRIAL: NCT04359966
Title: Prospective Randomised Trial of First and Second Line Treatments of Helicobacter Pylori Infection in Slovenia
Brief Title: Prospective Randomised Trial of First and Second Line Treatments of RCT of First and Second Line H Pylori Treatments in Slovenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Slovenian Society for Gastroenterology and Hepatology (Other)
Collaborators: KRKA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZGH Krka
Record Dates: First submitted 2020-04-17; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Helicobacter Pylori Infection; Eradication Treatments
Keywords: Helicobacter pylori; First line treatment; Second line treatment; susceptibility to antibiotics
MeSH Terms: interventions — Esomeprazole; Clarithromycin; Metronidazole; bismuth tripotassium dicitrate; Amoxicillin; Levofloxacin; Ofloxacin

STUDY DESIGN:
Intervention Model Description: Randomised procpective multicenter trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- First line therapy for H pylori infection (Active Comparator): Tripple 14 day first line therapy Esomeprazole 40 mg, Clarithromycin 500 mg, Amoxicillin 1000 mg, all BID 14 days
  Interventions: Drug: Esomeprazole 40mg, Clarithromycin 500 mg, Metronidazole 400 mg,
- First line therapy for H pylori infection second arm (Experimental): Bismuth quadruple first line therapy
  Bismuth subcitrat 120 mg , Amoxicillin 500 mg, Metronidazole 400 mg, all QID, Esomeprazole 40 mg BID, 14 days.
  Interventions: Drug: Esomeprazole 40mg, Bismuth subcitrate 120 mg, Amoxicillin 500 mg, Metronidazole 400 mg
- Second line therapy for H pylori infection (Active Comparator): Bismuth quadruple second line therapy for those treated with Tripple first line therapy
  Bismuth subcitrat 120 mg , Amoxicillin 500 mg, Metronidazole 400 mg, all QID, Esomeprazole 40 mg BID, 14 days.
  Interventions: Drug: Esomeprazole 40mg, Bismuth subcitrate 120 mg, Amoxicillin 500 mg, Metronidazole 400 mg
- Second line therapy for H pylori infection second arm (Experimental): Tripple second line therapy
  Esomeprazol 40 mg BID Amoxicillin 1000 mg BID, Levofloxacin 500 mg OID, 14 days or
  Interventions: Drug: Esomeprazole 40mg, Amoxicillin 500 mg, Levofloxacin 500 mg

INTERVENTIONS:
Drug: Esomeprazole 40mg, Clarithromycin 500 mg, Metronidazole 400 mg, — First line therapy
  Other Names: Emozul, Fromilid,Efloran
  Arms: First line therapy for H pylori infection
Drug: Esomeprazole 40mg, Bismuth subcitrate 120 mg, Amoxicillin 500 mg, Metronidazole 400 mg — First line therapy second arm
  Other Names: Emozul, Bismut oksid Krka, Hiconcil, Efloran
  Arms: First line therapy for H pylori infection second arm
Drug: Esomeprazole 40mg, Bismuth subcitrate 120 mg, Amoxicillin 500 mg, Metronidazole 400 mg — Second line therapy for Helicobacter pylori infection
  Other Names: Emozul, Bismut oksid Krka, Hiconcil, Efloran
  Arms: Second line therapy for H pylori infection
Drug: Esomeprazole 40mg, Amoxicillin 500 mg, Levofloxacin 500 mg — Second line therapy for Helicobacter pylori infection second arm
  Other Names: Emozul, Hiconcil,Tavanic
  Arms: Second line therapy for H pylori infection second arm

SUMMARY:
Study is prospective randomised multicentric. The primary objective of the study is to compare the efficacy of two first-line therapy regimens and two second-line therapy regimens (ie, after failure of first-line treatment) in patients with H. pylori infection. The secondary objective of the study is to determine the primary resistance of H. pylori to antibiotics in Slovenia.

DETAILED DESCRIPTION:
The infection with Helicobacter pylori is extremely widespread, as 60% of the world's population is infected. In Slovenia, the average prevalence is 25.1 %, the prevalence in the 20-year age group is 20 % and 76 % in patients in age group 50 - 75 years. All infected patients have active chronic gastritis, which is asymptomatic in most cases. Ulcers in the stomach or duodenum occurs in 15 % of patients. Due to chronic infection, MALT lymphoma or gastric cancer develop in 1 - 3 % of patients. According to the recommendations of the Slovenian Association for Gastroenterology and Hepatology, as well as European and other recommendations, everyone who is infected with Helicobacter pylori should be treated. H. pylori is a first-class carcinogen and is responsible for 50 % of all chronic cancer-causing infections in the developed world. Therefore, it is necessary to start programs of primary and secondary prevention of gastric cancer by searching and treating infected patients.

Patients infected with H. pylori who have not yet been treated will be randomly assigned to two first-line treatment groups:

Group 1: Esomeprazole 40 mg, Clarithromycin 500 mg, Amoxicillin 1000 mg, all BID,14 days Group 2: Bismuth subcitrate 120 mg, Amoxicillin 500 mg, Metronidazole 400 mg, all QID Esomeprazole 40 mg BID, 14 days

Patients unsuccessfully treated with first-line therapy will be randomly assigned to two second-line treatment groups:

Group 1: Esomeprazole 40 mg BID, Levofloxacin 500 mg OID, Amoxicillin 1000 mg BID, 14 days Group 2: Bismuth subcitrate 120 mg, Amoxicillin 500 mg, Metronidazole 400 mg, all QID, Esomeprazole 40 mg BID, 14 days

Inclusion criteria :

Patients 18 to 80 years of age. Patients have not received proton pump inhibitors for the past 14 days. Patients did not receive antibiotics last month. Helicobacter pylori infection has been demonstrated by rapid urease test

Exclusion criteria :

Prior treatment for Helicobacter pylori infection (in patients who will receive Schedule 1 eradication therapy).

Defects in blood clotting. taking anticoagulant medicines that make it impossible to take biopsies.

Drug allergy used in the study. Pregnancy, breastfeeding. Psychiatric illness that would prevent research participation. Active treatment for malignancy.

Statistical analysis:

To describe the variables, we will use the average value and standard deviation for the symmetrically distributed variables or median and 25th and 75th percentiles for asymmetrically distributed variables. Investigators will use the t-test for dependent variables or, in the case of asymmetrically distributed variables, the Wilcoxon test. To determine the differences between the two groups (Group 1 and Group 2) of the subjects, t-test for independent samples Will be used, or in the case of an asymmetrically distributed variables Mann-Whitney test.

ELIGIBILITY:
Inclusion criteria:

* Patients 18 to 80 years of age.
* Patients have not received proton pump inhibitors for the past 14 days.
* Patients did not receive antibiotics in the last month.
* Helicobacter pylori infection has been demonstrated by rapid urease test.

Exclusion Criteria:

* Prior treatment for Helicobacter pylori infection (in patients who will receive Schedule 1 eradication therapy).•
* Defects in blood clotting. taking anticoagulant medicines that make it impossible to take biopsies.
* Allergy to drugs used in the study.
* Pregnancy, breastfeeding shold be excluded.
* Psychiatric illness that would prevent research participation.
* Active treatment for malignancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2020-05-10 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Success rate of first line therapy for Helicobacter pylori infection | 2 years
  Eradication rate
Success rate of second line therapy for Helicobacter pylori infection | 3 years
  Eradication rate

SECONDARY OUTCOMES:
Helicobacter pylori resistance rate to antibiotics | 3 years
  Culture and susceptibility testing

CONTACTS AND LOCATIONS:
Overall Officials: BOJAN TEPES, Principal Investigator — AM DC Rogaška
Locations (3):
- Slovenia (3):
  - DC BLED, Bled
  - UCC, Ljubljana
  - Am Dc Rogaska, Rogaška Slatina

IPD SHARING:
Plan to Share IPD: No